CLINICAL TRIAL: NCT04464837
Title: Efficacy and Safety of Cold Snare Polypectomy (CSP) of Intermediate Sized Colorectal Polyps 10-15 mm With a Newly Designed Polypectomy Snare - A Feasibility Trial
Brief Title: Efficacy and Safety of Cold Snare Polypectomy (CSP) of Intermediate Sized Colorectal Polyps 10-15 mm
Acronym: COLDSNAP-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Monther Bajbouj, Principal Investigator, Technical University of Munich
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COLDSNAP-1
Record Dates: First submitted 2020-06-11; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Polyp; Colorectal Adenoma
Keywords: coldsnare polypectomy; hotsnare polypectomy; intermediate sized polyps

STUDY DESIGN:
Intervention Model Description: Proof-Of-Concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cold Snare Polypectomy of intermediate sized polyps (10-15 mm) — If an eligible polyp (10-15mm) is found, cold snare polypectomy is performed with the Olympus SnareMaster® Plus Snare
  Other Names: Olympus SnareMaster® Plus

SUMMARY:
Colorectal cancer (CRC) has become the third most common malignant tumor and is the second leading cause of cancer related deaths worldwide. Adenomatous polyps of the colon are possible precursor lesions for CRC. Screening for CRC has been shown effective in preventing CRC and related deaths, especially colonoscopy and resection of adenomatous polyps. Currently, for intermediate sized polyps 5 - 20 mm hot snare polypectomy (HSP) with the use of electrocautery is conventionally used, causing relevant adverse events including haemorrhage and postpolypectomy coagulation syndrome, but is safe regarding complete resection of the polyp due to burning effect on residual tissue. On the other hand, cold snare polypectomy (CSP) has grown popularity. Absence of electrocautery makes it technically easier and most important reduces adverse events. CSP is recommended as the preferred technique for polyps <5 mm by the European Society of Gastrointestinal Endoscopy (ESGE) guidelines. In literature, there is one multicenter trial from Japan recommending CSP for polyps 4-9 mm (average polyp size 5,4 mm) and only a few case studies for polyps 10-15 mm with inconsistent results, especially regarding the complete resection and pathological evaluation of the specimen.

In this feasibility trial, the investigators try to find out if CSP with a new designed polypectomy snare is efficient and safe in terms of complete resection (R0), pathological evaluation and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy
* signed informed consent
* at least one polyp of the size 10-15mm
* American Society of Anesthesiologists-classification (ASA) I-III

Exclusion Criteria:

* American Society of Anesthesiologists-classification (ASA) IV-VI
* Inflammatory bowel disease (IBD)
* known/suspected invasive colorectal cancer
* contraindications for polypectomy
* emergency indication for colonoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete Resection Rate (R0-resection) | 6 month
  Complete resection rate of polyps resected by cold snare polypectomy

SECONDARY OUTCOMES:
Required additional attempts for complete resection during surgery | during surgery
  Where there more than one attempts for complete resection of the polyp during surgery?
Incidence of immediate and delayed bleeding. | 3 weeks
  Immediate bleeding: Bleeding >30 seconds after snaring. Delayed bleeding: Bleeding during the next 3 weeks.
Technical Impossibility of CSP during surgery | during surgery
  Necessity of changing to HSP, if CSP is technically not possible

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Medical Department, Klinikum rechts der Isar, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ulrich JD, Rechberger P, Bachmann J, Herner A, V Figura G, Lahmer T, Phillip V, Mayr U, Haller B, Jesinghaus M, Schmid RM, Abdelhafez M, Schlag C. Efficacy and Safety of Cold Snare Polypectomy of Colorectal Polyps 10-15 mm with a Hybrid Snare: A Prospective Observational Pilot Study. Digestion. 2023;104(5):391-399. doi: 10.1159/000530642. Epub 2023 Jun 16. PMID 37331350